CLINICAL TRIAL: NCT02127086
Title: Managing Acute Pain in Critically Ill Non-communicative Palliative Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Virginia Commonwealth University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Carl Shanholtz, Associate Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HP-00053272; 4R01NR013664-04 (NIH)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Critically Ill
Keywords: Acute pain severity; Non-communicative patients; PAIN algorithm; Multi-dimensional Pain Assessment Tool (MOPAT)
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): The study design is a non-randomized quasi-experimental cohort design with two cohorts who will be sequentially studied. In phase 1, patients will comprise the usual care group (UCG), or control cohort, defined as receiving pain assessment and management practices that nurses are currently performing on the study units. In phase 2 the PAIN Algorithm coupled with analgesic order sets will be introduced to nurses and physicians on all participating units as the intervention. Patients enrolled in this phase will be considered the intervention group (IG), also called the experimental cohort. Nurses will be enrolled from the participating inpatient units to provide data on the clinical utility of the PAIN Algorithm.
  Interventions: Other: Intervention Group
- Usual Care Group (No Intervention): The study design is a non-randomized quasi-experimental cohort design with two cohorts who will be sequentially studied. In phase 1, patients will comprise the usual care group (UCG), or control cohort, defined as receiving pain assessment and management practices that nurses are currently performing on the study units. In phase 2 the PAIN Algorithm coupled with analgesic order sets will be introduced to nurses and physicians on all participating units as the intervention. Patients enrolled in this phase will be considered the intervention group (IG), also called the experimental cohort. Nurses will be enrolled from the participating inpatient units to provide data on the clinical utility of the PAIN Algorithm

INTERVENTIONS:
Other: Intervention Group — The PAIN Algorithm and analgesic order sets to be used by nurses to assess and reassess pain and opioid-related side effects will include orders for: 1) managing pain based on MOPAT Behavioral Dimension cut scores, 2) pre-medication before painful procedures, 3) titration of drugs, and 4) managing major opioid side effects. The order sets will start with small doses of opioids that will be titrated upwards for peak analgesic effect and allow for adjustment for patient characteristics and type of pain while simultaneously monitoring for and treating side effects.
  Other Names: PAIN algorithm; Analgesic Order Set; Experimental Arm
  Arms: Intervention Group

SUMMARY:
The purpose of this project is to test an innovative method for managing pain in acutely ill hospitalized patients who are not able to report their pain verbally to health care professionals. Nurses will use a Pain Assessment and Intervention for the Non-communicative (PAIN) Algorithm to guide assessment of pain, selection of pain medications, and management of medication side effects. The researchers will evaluate whether patients who are managed with the PAIN Algorithm have less severe pain and increased use of pharmacologic pain management strategies than those who are not managed with the PAIN Algorithm.

The study design is a non-randomized quasi-experimental cohort design with two cohorts who will be sequentially studied. In phase 1, patients will comprise the usual care group (UCG), or control cohort, defined as receiving pain assessment and management practices that nurses are currently performing on the study units. In phase 2 the PAIN Algorithm coupled with analgesic order sets will be introduced to nurses and physicians on all participating units as the intervention. Patients enrolled in this phase will be considered the intervention group (IG), also called the experimental cohort. Nurses will be enrolled from the participating inpatient units to provide data on the clinical utility of the PAIN Algorithm

DETAILED DESCRIPTION:
The Multiple Principal Investigators (MPIs) are Dr. Deborah McGuire (VCU) and Dr. Carl Shanholtz (University of Maryland. University of Maryland Medical Center (UMMC) delivers palliative care to acutely ill persons across a range of ages, medical illnesses, and traumatic injuries for whom death is not a foregone conclusion. Data will be collected on eight inpatient acute care nursing units, which are grouped into services defined by medical specialties and patients: Medical Intensive Care Unit, Medical Intermediate Care Unit (IMC), Neuro-Trauma IMC Unit, Neuro-Trauma Critical Care Unit, Multi-trauma Critical Care Unit, Select Trauma IMC Unit, Select Trauma Critical Care, and Surgical Intensive Care Unit. Average lengths of stay are highly variable but are generally a week or less. This is a one site, quasi-experimental cohort control group design, conducted in two sequential phases with repeated measures in two different but comparable cohorts. The primary aim is to test whether a pain algorithm that incorporates the Multi-dimensional Pain Assessment Tool (MOPAT) and an analgesic order set improves pain severity and use of pharmacologic pain management strategies in critically ill non-communicative palliative care patients who are hospitalized on medical, surgical, and trauma intensive care units when compared to patients without the algorithm. The secondary descriptive aims are to: (S1) compare pain severity and use of pharmacologic pain management strategies in patients with and without concurrent pain-related conditions, (S2) describe the pattern of patients' pain over time, and (S3) evaluate nurses' perceptions of clinical utility of the pain algorithm. This study has two samples: non-communicative palliative care patients who have acute pain and nurses who will use the PAIN Algorithm and order set to manage their patients' pain. Patients will be 300 critically ill adults who are non-communicative for a variety of reasons (intubation, neurological impairment, etc.) and have conditions that are known to produce acute pain. Patient data collection will be collected for 7 days (day 1 to 7) or until the patient dies, regains the ability to self-report pain, is transferred to a non-participating unit, or is discharged, whichever comes first. This timeframe is based on average lengths of stay for non-communicative patients on the units, quality of care benchmarks for pain relief in self-reporting patients, and practical considerations for research in acutely ill individuals. Volunteer Staff Nurse data will be collected at baseline and monthly over 24-36 months. Study Phase 1 will occur before introduction of the pain algorithm which occurs in Phase 2. Prior to starting this phase, nurses will be trained to use the MOPAT and it will be incorporated into the pain standard of care and the electronic medical record (EMR), permitting comparison of pain assessment data between Phases 1 and 2. The MOPAT will replace the Checklist of Nonverbal Pain Indicators (CNPI), which is currently used to assess pain in non-communicative patients but has multiple limitations. Following a 6 week run-in period in which nurses' appropriate and universal use of the MOPAT is assessed and assured, data collection will begin. Patients in this cohort will comprise the usual care group (UCG), or control cohort. Nurses will also be enrolled from the participating inpatient units. Usual care is defined as all pain assessment and management practices that nurses are currently performing on the study units, including inconsistent use of existing algorithms and protocols. Data will be collected on patients and nurses until we accrue 150 patients. Study Phase 2 will begin following the completion of Phase 1. Prior to starting this phase, our pain algorithm, christened the Pain Assessment and Intervention for the Non-communicative (PAIN) Algorithm, will be introduced to nurses and physicians on all participating units and they will be trained in its use. The PAIN Algorithm couples the MOPAT with an analgesic order set. The final algorithm will have specific numerical cut points derived from a consensual process. In addition, orders in the order set, and adaptations to accommodate patient demographic and medical variables will be finalized through a detailed collaborative process. After a 6 week run-in period to assure appropriate use of the PAIN Algorithm, data collection will begin. Patients enrolled in phase 2 will be considered the intervention group (IG), also called the experimental cohort. We will collect the same patient and nurse data as in Phase 1, with the addition of nurse perceptions of clinical utility of the PAIN Algorithm, and will continue until we have accrued 150 patients. Considerations regarding potential risks to patients are as follows. Because the algorithm includes opioids, and patients targeted in this study will be critically ill with numerous pathological processes that could be adversely affected by these drugs, there is concern about adverse opioid-related side effects such as sedation and respiratory depression. To deal with this concern, the PAIN Algorithm order set will include orders for routine monitoring of these side effects and interventions to manage them, for example, titrating the opioid dose or using a reversing agent in the case of severe respiratory depression. To ensure that these orders conform to standards for safe practice, the interdisciplinary panel that develops the analgesic order set in conjunction with the researchers will build in drug side effect assessment, treatment, and reassessment. Another area of potential risk, however, remains of concern. Since the MOPAT instrument is a relatively new pain assessment tool, and medication decisions will be made using MOPAT Behavioral Dimension scores, there is the possibility that treatment decision may under-medicate, or overmedicate a patient's pain. Thus, even with careful attention to drug side effects, the study is probably greater than minimal risk. There are no alternative treatments and procedures, since the PAIN Algorithm will be integrated into clinical practice as the standard of care while the patient is on study. There are no anticipated potential risks to the volunteer study nurses who consent to participate in the study. Since the PAIN Algorithm with the analgesic order set will be incorporated into standard of care all nurses on the inpatient units will use it whether or not they consent to participate in the study. Those nurses who consent will provide demographic and practice data, and provide monthly appraisals of usefulness of the MOPAT in Phase 1, and the PAIN Algorithm (including MOPAT) in Phase 2 and will not be affected by the study intervention. Because there is always a risk of opioid-induced side effects when opioids are used to manage pain, the PAIN Algorithm analgesic order set includes provisions for monitoring, detecting, and managing such side effects thus making the algorithm potentially safer than usual care which does not generally include side effect monitoring. There are no physical or psychosocial risks to nurses who consent to participate in the study. For both patient and nurse subjects, protection of confidentiality is a concern. Therefore, all patient and nurse data collection forms will contain only the unique study identification numbers, with the master list kept in a locked file cabinet in a locked project office. When the study is completed, the list will be destroyed and all data will be identified only by study identification numbers. Only the PI and project manager will have access to these lists during the study. Standard operating procedures for analysis activities, such as recruitment, data collection, data management, data analysis, reporting of adverse events, and change in management are outlined in the study manual of operating procedures. Source data include: electronic medical records, patient's paper charts, data collection "teleforms" . The manual of operations also includes standard operating procedures for data entry, transfer, and quality assurance. "Teleforms" have a built in quality checks including predetermined rules for range and consistency with other study data fields. The plan for statistical analysis is as follows.The primary aim testing that there is a decrease in pain severity for the intervention group as compared to the usual care group, will use the interaction F-test from 2 x 4 repeated measures analysis. If test assumptions are not met, or if there is missing data, mixed linear modeling will be used that does not require sphericity or complete data. Specific comparisons also will be made between the groups at both 2 and 4 days using interaction contrasts. The number and total dosage of pharmacologic interventions will be computed for each time period using the American Pain Society equi-analgesic table.To test for an increase in the number of pharmacologic agents used for pain and an increase in the total equi-analgesic dosage of pharmacologic agents used for pain a 2 X 3 ANOVA or mixed linear modeling approach will be used depending on whether assumptions are met. To address covariates and control for unit-based effects, first a comparison of units to identify unit-level differences, such as type of service or ambient environment, that might be related to patient outcomes and then include them in a hierarchical linear model will be conducted. Patient demographic variables such as age and gender and clinical variables such as pain-related conditions, type of pain and co-analgesics, and Glasgow Coma Scale score will be examined for their relationship to outcomes and incorporated as factors or covariates depending on the level of measure and strength of bivariate relationship. These variables can be incorporated into a hierarchical model or, if unit-level differences are not relevant, then into analysis of covariance or multiple regression models. The secondary aims will be analyzed using descriptive approaches. For (S1) patients will be categorized on the basis of whether they have pain-related conditions using the Clinical Classification System and a 2 x 4 repeated measures analysis will be used to compare these two groups on pain severity and a 2 x 3 repeated measures analysis to compare the number and types of drug categories and total dosage of pharmacologic agents. If there is a significant interaction effect, the groups will be compare at each time point as post-hoc analyses. For (S2) a descriptive pattern of patients' pain over time will be examined. Of interest is whether there are sub-groups of patients who demonstrate different patterns. A graphic techniques (e.g., spaghetti plots) will be used to identify sub-groups and attempt to describe them based on clinical and demographic variables. In addition, we will compute the change in pain between the time periods and plot the cumulative distribution function at each time point as an initial step in identifying potential cut points to define a clinical important change. To evaluate nurse perceptions of the clinical utility of the PAIN Algorithm and the MOPAT (S3), we will examine the frequency distribution for responses to each item on the Clinical Utility Questionnaire (CUQ) and the overall summated response. For CUQ items that are used in evaluating MOPAT utility in both phases, the responses will be compared using t-tests. In addition, the percentage of nurses who agree or strongly agree with each statement and make comparisons based on nurse demographic and practice characteristics will be done.

ELIGIBILITY:
Inclusion Criteria Patients:

* 18 years of age or older
* Diagnosed with potentially life-threatening conditions accompanied by acute pain
* With or without concurrent pain-related conditions
* Unable to self-report pain
* Receiving care on the participating units

Exclusion Criteria Patients:

* Receiving paralytic agents
* Sedated and with a Richmond Agitation Sedation Scale score of -5
* Able to communicate pain through any verbal or physical means such as nodding or wiggling fingers

Inclusion Criteria Nurses:

* Assigned to a participating unit
* Working at least 36 hours/week

Exclusion Criteria Nurses:

* Routinely rotating between participating and non-participating units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2015-03; Primary Completion 2017-06-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Acute pain severity (patient outcome variable) | Acute pain severity measured with same tool daily for 7 days
  Is measured using: (1) Multi-dimensional Objective Pain Assessment Tool (MOPAT) a measure of acute pain severity consisting of two dimensions -Behavioral Dimension of four items scored from 0-3 depending on severity and Physiologic Dimension of four items scored as no change or change from usual. Because the Physiologic Dimension has lower reliability and literature indicating that physiologic indicators are not consistent measures of acute pain, only the Behavioral Dimension scores is to make decisions about orders in the analgesic order set.

SECONDARY OUTCOMES:
Use of pharmacologic pain management strategies (patient outcome variable) | electronic health record data downloaded from each patient record after completing 7 days on study
  Pain management data charted by the nurses caring for patients in Phases 1 and 2 will be downloaded from the electrical health record into an Excel data file. These data are based on a clinical dataset and methods routinely used to monitor pain management and quality. These data include total amount of opioids administered, categorized into as needed (PRN) and scheduled drugs, and converted into morphine equivalents.

OTHER OUTCOMES:
Clinical utility (nurse outcome variable) | 32 months
  Clinical Utility is defined as the usefulness of a measure or an algorithm within a specific setting and clinical population including the extent to which it can be used by practicing nurses. In study phase 1 the clinical utility of the Multi-dimensional Pain Assessment Tool (MOPAT) and in study phase 2 measures the clinical utility of the PAIN Algorithm, including the analgesic order set, by adding items that appraise the algorithm and order set in terms of ease of use, guidance in managing pain, etc.
Patterns of pain (patient outcome variable) | 7 days
  The patterns of each patient's pain will be categorized by abstracting MOPAT scores from the Electronic Medical Record(EMR) and entering the data into an excel file, and analyzing using graphic techniques.
Concurrent pain related conditions (patient outcome variable) | 7 days
  Each patient's concurrent pain related conditions will be abstracted from the Electronic Medical Record (EMR).

CONTACTS AND LOCATIONS:
Overall Officials: Carl Shanholtz, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Acute Pain Management Guideline Panel. Acute pain management: operative or medical procedures and trauma. Clinical practice guideline Publ No. 92-0032. Rockville, MD: Agency for Health Care Policy and Research, Public Health Service, U.S. Department of Health and Human Services; 1992.
- [Background] Ahles TA, Ruckdeschel JC, Blanchard EB. Cancer-related pain--II. Assessment with visual analogue scales. J Psychosom Res. 1984;28(2):121-4. doi: 10.1016/0022-3999(84)90004-7. PMID 6737324
- [Background] Anderson F, Downing GM, Hill J, Casorso L, Lerch N. Palliative performance scale (PPS): a new tool. J Palliat Care. 1996 Spring;12(1):5-11. PMID 8857241
- [Background] Arbour C, Gelinas C. Are vital signs valid indicators for the assessment of pain in postoperative cardiac surgery ICU adults? Intensive Crit Care Nurs. 2010 Apr;26(2):83-90. doi: 10.1016/j.iccn.2009.11.003. Epub 2009 Dec 30. PMID 20044256
- [Background] Bailey FA, Burgio KL, Woodby LL, Williams BR, Redden DT, Kovac SH, Durham RM, Goode PS. Improving processes of hospital care during the last hours of life. Arch Intern Med. 2005 Aug 8-22;165(15):1722-7. doi: 10.1001/archinte.165.15.1722. PMID 16087819
- [Background] Bausell RB, Li Y. Power analysis for experimental research. Cambridge, England: Cambridge University Press; 2002.
- [Background] Bertsche T, Askoxylakis V, Habl G, Laidig F, Kaltschmidt J, Schmitt SP, Ghaderi H, Bois AZ, Milker-Zabel S, Debus J, Bardenheuer HJ, Haefeli WE. Multidisciplinary pain management based on a computerized clinical decision support system in cancer pain patients. Pain. 2009 Dec 15;147(1-3):20-8. doi: 10.1016/j.pain.2009.07.009. Epub 2009 Aug 19. PMID 19695779
- [Background] Botti M, Bucknall T, Manias E. The problem of postoperative pain: issues for future research. Int J Nurs Pract. 2004 Dec;10(6):257-63. doi: 10.1111/j.1440-172x.2004.00487.x. PMID 15544581
- [Background] Cade CH. Clinical tools for the assessment of pain in sedated critically ill adults. Nurs Crit Care. 2008 Nov-Dec;13(6):288-97. doi: 10.1111/j.1478-5153.2008.00294.x. PMID 19128312
- [Background] Caraceni A, Cherny N, Fainsinger R, Kaasa S, Poulain P, Radbruch L, De Conno F. Pain measurement tools and methods in clinical research in palliative care: recommendations of an Expert Working Group of the European Association of Palliative Care. J Pain Symptom Manage. 2002 Mar;23(3):239-55. doi: 10.1016/s0885-3924(01)00409-2. PMID 11888722
- [Background] Chanques G, Jaber S, Barbotte E, Violet S, Sebbane M, Perrigault PF, Mann C, Lefrant JY, Eledjam JJ. Impact of systematic evaluation of pain and agitation in an intensive care unit. Crit Care Med. 2006 Jun;34(6):1691-9. doi: 10.1097/01.CCM.0000218416.62457.56. PMID 16625136
- [Background] Cohen SP, Christo PJ, Moroz L. Pain management in trauma patients. Am J Phys Med Rehabil. 2004 Feb;83(2):142-61. doi: 10.1097/01.PHM.0000107499.24698.CA. PMID 14758300
- [Background] Downing,MG. Palliative Performance Scale (PPSv3) version 2. Learning Center for Palliative Care. Victoria, BC. 2005.
- [Background] Perreault SD. Chromatin remodeling in mammalian zygotes. Mutat Res. 1992 Dec;296(1-2):43-55. doi: 10.1016/0165-1110(92)90031-4. PMID 1279407
- [Background] Foley K. Acute and chronic cancer pain syndromes. Chapter 8.2.2. In: Doyle D, Hanks G, Cherney NI, Calman K, eds. Oxford Textbook of Palliative Medicine 3rd ed. New York, NY: Oxford University Press 298-316, 2005.
- [Background] Gil Z, Smith DB, Marouani N, Khafif A, Fliss DM. Treatment of pain after head and neck surgeries: control of acute pain after head and neck oncological surgeries. Otolaryngol Head Neck Surg. 2006 Aug;135(2):182-8. doi: 10.1016/j.otohns.2006.03.005. PMID 16890065
- [Background] Health Care Cost and Utilization Project (HCUP). Clinical Classifications Software (CCS) for ICD-9-CM. http://www.hcup-us.ahrq.gov/toolssoftware/ccs/ccs.jsp#overview. Updated Jan 25, 2011. Accessed March 20, 2011.
- [Background] Herr K, Bjoro K, Decker S. Tools for assessment of pain in nonverbal older adults with dementia: a state-of-the-science review. J Pain Symptom Manage. 2006 Feb;31(2):170-92. doi: 10.1016/j.jpainsymman.2005.07.001. PMID 16488350
- [Background] Herr K, Coyne PJ, Key T, Manworren R, McCaffery M, Merkel S, Pelosi-Kelly J, Wild L; American Society for Pain Management Nursing. Pain assessment in the nonverbal patient: position statement with clinical practice recommendations. Pain Manag Nurs. 2006 Jun;7(2):44-52. doi: 10.1016/j.pmn.2006.02.003. PMID 16730317
- [Background] Herr K, Titler M, Fine P, Sanders S, Cavanaugh J, Swegle J, Forcucci C, Tang X. Assessing and treating pain in hospices: current state of evidence-based practices. J Pain Symptom Manage. 2010 May;39(5):803-19. doi: 10.1016/j.jpainsymman.2009.09.025. PMID 20471542
- [Background] International Association for the Study of Pain (IASP) Task Force on Acute Pain. Management of Acute Pain: A Practical Guide. Ready LB, Edwards WT, eds. Seattle, Washington; IASP Publications; 1992.
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Johnston CC. Psychometric issues in the measurement of pain. In: Finley GA, McGrath PJ, eds. Measurement of Pain in Children and Infants. Seattle, WA: IASP Press 5-20, 1998.
- [Background] Kaiser K, Dupee J, Petri L, Hill J, Smith D. Application of selected 2008 American pain society quality indicators for acute and chronic pain. Journal of Pain 8(4):S1-S70, 2007.
- [Background] Kaiser K. Use of electronic medical records in pain management In: Pasero C, McCaffery M. Pain Assessment and Pharmacologic Management. Baltimore, MD: Mosby 837-857, 2011.
- [Background] Kessler SM, Swetz KM. Prognostication in severe traumatic brain injury in adults #239. J Palliat Med. 2011 Jun;14(6):782-3. doi: 10.1089/jpm.2011.9682. No abstract available. PMID 21651368
- [Background] Malchow RJ, Black IH. The evolution of pain management in the critically ill trauma patient: Emerging concepts from the global war on terrorism. Crit Care Med. 2008 Jul;36(7 Suppl):S346-57. doi: 10.1097/CCM.0b013e31817e2fc9. PMID 18594262
- [Background] Melzack R, Casey KL. Sensory, Motivational, and Central Control Determinants of Pain: A New Conceptual Model. Kenshalo D. (Ed.). Chas C. Thomas. Springfield, MA; 423-439, 1968.
- [Background] . McGuire DB. The multidimensional phenomenon of cancer pain. In: McGuire DB, Yarbro CH, eds. Cancer Pain Management. Orlando, FL: Grune and Stratton 1-20, 1987.
- [Background] McGuire DB, Ahles TA, Dudley WN, Yeager KA. Multidimensional conceptualization of acute oral pain in transplant and leukemia patients. Psycho-Oncology 8:6S23, 1999.
- [Background] McGuire DB, DeLoney VG, Yeager KA, Owen DC, Peterson DE, Lin LS, Webster J. Maintaining study validity in a changing clinical environment. Nurs Res. 2000 Jul-Aug;49(4):231-5. doi: 10.1097/00006199-200007000-00007. PMID 10929695
- [Background] McGuire DB. The multiple dimensions of cancer pain: a framework for assessment and management. In: McGuire DB, Yarbro CH, Ferrell BR, eds. Cancer Pain Management 2nd ed. Boston, MA: Jones and Bartlett Publishers; 1-17: 1995.
- [Background] McGuire DB. Occurrence of cancer pain. J Natl Cancer Inst Monogr. 2004;(32):51-6. doi: 10.1093/jncimonographs/lgh015. PMID 15263041
- [Background] McGuire DB, Kaiser K, Soeken K, Reifsnyder J, Keay T. Measuring pain in noncommunicative palliative care patients in the acute care setting: Psychometric evaluation of the multidimensional objective pain assessment tool (MOPAT). Journal of Pain and Symptom Management 41(1):299-300, 2011.
- [Background] Mercadante S, Radbruch L, Caraceni A, Cherny N, Kaasa S, Nauck F, Ripamonti C, De Conno F; Steering Committee of the European Association for Palliative Care (EAPC) Research Network. Episodic (breakthrough) pain: consensus conference of an expert working group of the European Association for Palliative Care. Cancer. 2002 Feb 1;94(3):832-9. doi: 10.1002/cncr.10249. PMID 11857319
- [Background] Mularski RA, Curtis JR, Billings JA, Burt R, Byock I, Fuhrman C, Mosenthal AC, Medina J, Ray DE, Rubenfeld GD, Schneiderman LJ, Treece PD, Truog RD, Levy MM. Proposed quality measures for palliative care in the critically ill: a consensus from the Robert Wood Johnson Foundation Critical Care Workgroup. Crit Care Med. 2006 Nov;34(11 Suppl):S404-11. doi: 10.1097/01.CCM.0000242910.00801.53. PMID 17057606
- [Background] National Consensus Project for Quality Palliative Care (NCP). Clinical Practice Guidelines for Quality Palliative Care (2nd ed.). Brooklyn, NY: Author; 2009.
- [Background] National Institute of Nursing Priority Expert Panel on Symptom Management: Acute Pain. 6. Symptom Management: Acute Pain. National Institute of Health Nursing Research, U.S. Department of Health and Human Services, U.S. Public Health Service, National Institutes of Health. Bethesda, MD: NIH Pub. No 94-24211; 1994.
- [Background] National Priorities Partnership (NPP). National Priorities and Goals: Aligning our Efforts to Transform America's Healthcare. Washington, DC: National Quality Forum; 2008.
- [Background] National Quality Forum (NQF). A National Framework and Preferred Practices for Palliative and Hospice Care Quality. Washington DC: Author; 2006.
- [Background] Paice JA, Muir JC, Shott S. Palliative care at the end of life: comparing quality in diverse settings. Am J Hosp Palliat Care. 2004 Jan-Feb;21(1):19-27. doi: 10.1177/104990910402100107. PMID 14748519
- [Background] Prescott PA, Soeken KL. The potential uses of pilot work. Nurs Res. 1989 Jan-Feb;38(1):60-2. doi: 10.1097/00006199-198901000-00015. No abstract available. PMID 2911515
- [Background] Resnick B, Inguito P, Orwig D, Yahiro JY, Hawkes W, Werner M, Zimmerman S, Magaziner J. Treatment fidelity in behavior change research: a case example. Nurs Res. 2005 Mar-Apr;54(2):139-43. doi: 10.1097/00006199-200503000-00010. PMID 15778656
- [Background] Reyna YZ, Bennett MI, Bruera E. Ethical and practical issues in designing and conducting clinical trials in palliative care. In: Addington-Hall JM, Bruera E, Higginson IJ, Payne S, eds. Research Methods in Palliative Care. New York, NY: Oxford; 27-38, 2009.
- [Background] Reynolds CM, Suber F, Curtis KM, Henriques HF. A novel pain management protocol results in more rapid analgesia for trauma patients. Society for Academy of Emergency Medicine 11(5):497, 2004.
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Sessler CN, Grap MJ, Ramsay MA. Evaluating and monitoring analgesia and sedation in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S2. doi: 10.1186/cc6148. Epub 2008 May 14. PMID 18495053
- [Background] . Shadish WR, Cook TD, Campbell DT. Experimental and Quasi-experimental Designs for Generalized Causal Inference. Belmont, CA: Wadsworth; 2002.
- [Background] Strickland OL, Jackson G, Gilead M, McGuire DB, Quarles S. Use of focus groups for pain and quality of life assessment in adults with sickle cell disease. J Natl Black Nurses Assoc. 2001 Dec;12(2):36-43. PMID 11902019
- [Background] van Eyk HG, Terhorst C, de Vijlder MM. Fragmentation of human IgG globulin with papain, trypsin and pepsin. Clin Chim Acta. 1967 Jun;16(3):429-31. doi: 10.1016/0009-8981(67)90309-9. No abstract available. PMID 4166544
- [Background] Teasdale G, Murray G, Parker L, Jennett B. Adding up the Glasgow Coma Score. Acta Neurochir Suppl (Wien). 1979;28(1):13-6. doi: 10.1007/978-3-7091-4088-8_2. No abstract available. PMID 290137
- [Background] Truog RD, Campbell ML, Curtis JR, Haas CE, Luce JM, Rubenfeld GD, Rushton CH, Kaufman DC; American Academy of Critical Care Medicine. Recommendations for end-of-life care in the intensive care unit: a consensus statement by the American College [corrected] of Critical Care Medicine. Crit Care Med. 2008 Mar;36(3):953-63. doi: 10.1097/CCM.0B013E3181659096. PMID 18431285
- [Background] Twaddle ML, Maxwell TL, Cassel JB, Liao S, Coyne PJ, Usher BM, Amin A, Cuny J. Palliative care benchmarks from academic medical centers. J Palliat Med. 2007 Feb;10(1):86-98. doi: 10.1089/jpm.2006.0048. PMID 17298257
- [Background] Vallano A, Malouf J, Payrulet P, Banos JE; Catalan Research Group for the Study of Pain in the Hospital. Analgesic use and pain in the hospital settings. Eur J Clin Pharmacol. 2007 Jun;63(6):619-26. doi: 10.1007/s00228-007-0303-7. Epub 2007 Apr 20. PMID 17447056
- [Background] Virik K, Glare P. Validation of the palliative performance scale for inpatients admitted to a palliative care unit in Sydney, Australia. J Pain Symptom Manage. 2002 Jun;23(6):455-7. doi: 10.1016/s0885-3924(02)00407-4. No abstract available. PMID 12067769
- [Background] Walker KA, Nachreiner D, Patel J, Mayo RL, Kearney CD. Impact of standardized palliative care order set on end-of-life care in a community teaching hospital. J Palliat Med. 2011 Mar;14(3):281-6. doi: 10.1089/jpm.2010.0398. PMID 21361835
- [Background] Waltz CF, Strickland OL, Lenz ER. Measurement in Nursing Research. Philadelphia, PA: FA Davis; 1984.